CLINICAL TRIAL: NCT06620705
Title: Pacing Away from Heart Failure: Left Bundle Branch Area Pacing or Biventricular Pacing in Patients with Atrial Fibrillation and Left Ventricular Dysfunction
Brief Title: Left Bundle Branch Area Pacing or Biventricular Pacing in AF and Left Ventricular Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: srdpiers (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, srdpiers, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL84372.058.23
Record Dates: First submitted 2024-09-10; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Block, Heart; Pacing-Induced Cardiomyopathy
Keywords: pacing; cardiac resynchronization therapy; left bundle branch area pacing; conduction system pacing; heart failure; heart block
MeSH Terms: conditions — Heart Failure; Heart Block | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Randomized patient and assessor blinded non-inferiority cross-over trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to the treatment allocation. The assessor of the ECG endpoints and echocardiographic endpoints will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left bundle branch area pacing (Experimental): 6 months of left bundle branch area pacing.
  Interventions: Device: Left bundle branch area pacing
- Biventricular pacing (Active Comparator): 6 months of biventricular pacing using a RV apex lead and LV lead in the coronary sinus.
  Interventions: Device: Biventricular pacing

INTERVENTIONS:
Device: Left bundle branch area pacing — Pacing of the left bundle branch area using a transvenous pacemaker lead
  Other Names: Conduction system pacing; Cardiac resynchronization therapy
  Arms: Left bundle branch area pacing
Device: Biventricular pacing — Pacing of the right and left ventricle using transvenous pacemaker leads
  Other Names: Cardiac resynchronization therapy
  Arms: Biventricular pacing

SUMMARY:
It is unknown whether left bundle branch area pacing (LBBAP) or biventricular pacing best prevents or reverses left ventricular (LV) adverse remodelling in patients with atrial fibrillation (AF) who require ventricular pacing or CRT. This randomized non-inferiority cross-over trial will compare left ventricular end-systolic volume change and secondary endpoints between LBBAP and biventricular pacing in patients with AF and LV dysfunction.

DETAILED DESCRIPTION:
Rationale: Patients with atrial fibrillation (AF) and left ventricular (LV) dysfunction may require ventricular pacing because of bradycardia, AV junction ablation, or for cardiac resynchronization therapy. Right ventricular (RV) pacing is associated with the risk of adverse LV remodelling and heart failure, in particular in those with pre-existing LV dysfunction. Both LBBAP and biventricular pacing can prevent LV dyssynchrony. It is unknown which pacing mode best prevents or reverses LV adverse remodelling in patients with AF who require ventricular pacing or CRT.

Primary objectives:

1. To compare LVESV change between LBBAP and biventricular pacing in patients with AF and LV dysfunction.

   Secondary objectives:
2. To compare change in quality of life, New York Heart Association functional class, 6-minute walking distance, QRS duration, vectorcardiographic QRS area, left ventricular ejection fraction (LVEF), global longitudinal strain and NT-proBNP between LBBAP and biventricular pacing in patients with AF and LV dysfunction.

Study design: Randomized patient and assessor blinded non-inferiority cross-over trial.

Study population: Patients with permanent AF and LVEF < 50% who require ventricular pacing because of bradycardia, AV junction ablation, or CRT.

Intervention: Patients will be randomized according to a crossover design to first 6 months of LBBAP and then 6 months of biventricular pacing, or vice versa.

After finishing the randomization phase of the study at 12 months, patients will be followed according to routine clinical practice. Clinical follow-up, an ECG, device interrogation and echocardiography will be performed at 36 months (2 years after finishing the randomization phase) in all patients.

Main study parameters/endpoints: New York Heart Association (NYHA) functional class, Minnesota Living with Heart Failure Questionnaire (MLHFQ), 6-minute walking distance, ECG (vectorcardiographic QRS area, QRS duration), echocardiography (LVESV, LVEF, global longitudinal strain), NT-proBNP, lead and device performance (sensing, pacing, expected battery life), complications and costs will be evaluated for each pacing mode.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For the purpose of this randomized controlled trial, patients will also receive a LBBAP lead. The additional risk of serious adverse events is ~1.5% (lead dislodgement 1.1%, 0.4% acute coronary syndrome [all managed conservatively without further sequelae in prior studies]).(1) Patients who participate in the trial will have 3 extra follow-up visits, 4 extra questionnaires, 3 extra ECGs, 3 extra device interrogations, 3 extra echocardiograms and 4 extra blood samples (5 mL each).

ELIGIBILITY:
INCLUSION CRITERIA

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Adults ≥18 years with permanent AF and LVEF < 50% who either require ventricular pacing because of bradycardia including patients undergoing AV junction ablation, or have an indication for cardiac resynchronization therapy.
* Expected percentage of ventricular pacing > 40%
* ≥ 3 months of heart failure medication optimization

Of note, patients who already have a device, but require an upgrade to a CRT device, can also be included

EXCLUSION CRITERIA

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Age < 18 years
* Pregnancy or active pregnancy wish
* Not eligible for implantation of an RV lead, LBBAP lead, or LV lead in the coronary sinus
* Recent valve intervention/surgery or acute myocardial infarction (< 6 months)
* NYHA functional class IV heart failure, left ventricular assist device or cardiac transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Left ventricular end-systolic volume (LVESV) change | 6 months
  Left ventricular end-systolic volume change measured by echocardiography

SECONDARY OUTCOMES:
Change in New York Heart Association functional class | 6 months
  Change in New York Heart Association functional class (NYHA)
Change in Minnesota living with heart failure questionnaire | 6 months
  The Minnesota living with heart failure questionnaire (MLHFQ) is a self-administered disease-specific questionnaire for patients with heart failure, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of heart failure on quality of life, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst quality of life).
Change in 6-minute walking distance | 6 months
  Change in 6-minute walking distance
Change in QRS duration | 6 months
  Change in QRS duration on the 12-lead ECG
Change in vectorcardiographic QRS area | 6 months
  Change in vectorcardiographic QRS area on the vectorcardiogram reconstructed from a regular 12-lead ECG
Change in left ventricular function | 6 months
  Change in left ventricular function ejection fraction and global longitudinal strain on echocardiography
Change in NT-proBNP | 6 months
  Change in NT-proBNP as a heart failure biomarker
Complications | 6 months
  Complications related to device and leads
Lead pacing thresholds | 6 months
  Lead pacing thresholds, expressed as volts at pulse width (e.g. 0.4 V @ 0.4 ms). A lower pacing threshold is better.
Costs | 6 months
  Costs related to the device and leads

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiaan Piers, MD, PhD, Principal Investigator — Leiden University Medical Center, Leiden, the Netherlands
Locations (2):
- Aarhus University Hospital, Aarhus N, Aarhus N, Denmark
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with other researchers whenever reasonable and of potential benefit for patients.
Supporting Information: Study Protocol, CSR
Time Frame: After completion of the study and publication, the data will be shared with other researchers whenever reasonable and of potential benefit for patients.
Access Criteria: Whenever reasonable and of potential benefit for patients.